CLINICAL TRIAL: NCT03650634
Title: Prevalence of Erupted Supernumerary Teeth Among a Group of Egyptian Children Aged From Six to Fifteen Years Old: a Cross Sectional Study
Brief Title: Prevalence of Erupted Supernumerary Teeth Among a Group of Egyptian Children Aged From Six to Fifteen Years Old
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Riham Ahmed El-Halafawey Anwar Emam, Master student in Cairo University ( principal Investigator), Cairo University
Other Study IDs: CEBD-CU-2018-08-16
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Supernumerary Teeth
Keywords: supernumerary tooth; hyperdontia; mesiodens; paramolar
MeSH Terms: conditions — Tooth, Supernumerary

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the prevalence of erupted supernumerary teeth among a group of Egyptian children aged from 6-15 years old attending the Outpatients' clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
* Clinical examination will be done for participants fulfilling the inclusion criteria after obtaining an informed consent from parents for acceptance of participation in the study after explaining the purpose of the study and the measures that will be held to the child.
* A custom made examination chart (Appendix 1) will be filled out, during face to face interview with the child and/or his parents, including: date, name, age, gender, address, medical history and previous dental treatment followed by clinical examination to detect the presence of supernumerary teeth.
* The presence of supernumerary teeth and its type and location will be recorded in the examination chart.
* Each child with supernumerary teeth will be given a letter, translated into Arabic, outlining his dental status to inform the parents about the condition and the need for treatment

Examination chart (Appendix 1 ):

Date :...................................................................

Personal information:

Name............................................. Age..........................................

Gender :.......................................... Address : ................................

Phone number : .................................................. Medical history: ......................................................... ..................................................................................

Previous dental history: ...........................................

......................................................................................

Clinical examination :

Supernumerary teeth: presence / absence Location : ........................................... Type :..................................................

ELIGIBILITY:
Inclusion Criteria:

* Positive patient and parent acceptance for participation in the study.
* Patients who are medically free from any systemic disease.
* Children aged from 6 to 15 years old.
* Both sexes will be included.

Exclusion Criteria:

* Uncooperative children.
* Handicapped children.
* Children who refuse to participate in the study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will be selected from the Outpatients' clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University according to the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 604 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
prevalence of supernumerary teeth | 6 months
  Measuring device: clinical examination. Measuring unit : binary (yes or/ no ).

CONTACTS AND LOCATIONS:
Overall Officials: Randa Youssef, Ass.prof., Study Director — Cairo University; Rasha Hatem, Lecturer, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt